CLINICAL TRIAL: NCT04317976
Title: Impact of Ultrasound Guidance on the Performance of Accurate Cricoid and Paralaryngeal Pressure
Brief Title: Ultrasound Guided Cricoid and Paralaryngeal Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Lim Siu Min, Dr,, University of Malaya
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2018118-6867; 45835 (Other: National Medical Research Register)
Record Dates: First submitted 2019-11-09; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Ultrasonography, Interventional
Keywords: Anatomy; oesophagus; ultrasound; incidence; cricoid; paralaryngeal

STUDY DESIGN:
Intervention Model Description: The study is a case-control intervention study, where all and every participant will be both the case and the control of their own.
Who Masked: Participant, Care Provider
Masking Description: Participant will not be informed of their anatomical details. Care provider will not be informed of their accuracy of performance of the airway manoeuvre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centrally located oesophagus post GA (Active Comparator): Oesophagus remained central after general anaesthesia, cricoid pressure applied by fingertips under ultrasound guidance
  Interventions: Other: cricoid pressure
- Eccentric located oesophagus post GA (Experimental): Oesophagus eccentric located after general anaesthesia, paralaryngeal pressure and cricoid pressure applied by fingertips under ultrasound guidance
  Interventions: Other: paralaryngeal pressure

INTERVENTIONS:
Other: paralaryngeal pressure — cricoid pressure with paralaryngeal pressure by fingertips applied under ultrasound guidance
  Arms: Eccentric located oesophagus post GA
Other: cricoid pressure — cricoid pressure by fingertips applied under ultrasound guidance
  Arms: Centrally located oesophagus post GA

SUMMARY:
The primary objective is to study impact of upper airway ultrasonography in guiding anaesthetic assistant into providing accurate cricoid pressure, or both cricoid and paralaryngeal pressure in those with oesophagus deviation, achieving sonographic proven oesophageal occlusion compared to those without ultrasound guidance.

DETAILED DESCRIPTION:
All patients consented for the study were having their airway examined via US. Cross sectional sonography of the airway was performed to determine the anatomic relationship of the oesophagus relative to the trachea:

1. before induction of anaesthesia
2. after GA before external airway pressure manoeuvre
3. after GA with external airway pressure manoeuvre.

US guided CP was applied on subjects with central oesophagus; CP and PLP were applied on subject with eccentric oesophagus anatomy.

PLP was performed by lateral compression on the eccentric oesophagus by fingertips under US guidance. To standardised the application of CP and PLP, only 2 well trained investigators were allowed to performed the CP and PLP, US scan on airway and patient recruitment. The conduct of trial involved 2 investigators where first investigator provide US scan, and second investigator provide compression of CP or PLP using fingertips guided by the instruction of first investigator.

ELIGIBILITY:
Inclusion Criteria:

Elective list Under general anaesthesia Not intubated prior to OT

Exclusion Criteria:

Below 18 years old Pregnant Neck deformities Previous maxillofacial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The number of patients with eccentric oesophagus under general anesthesia, successfully occluded by using cricoid and paralaryngeal pressure. | ultrasound assessment of oesophagus done after general anaesthesia, during application of cricoid pressure, and during application of cricoid and paralaryngeal pressure
  we are studying the effectiveness of cricoid pressure versus cricoid and paralaryngeal pressure(novel technique) in those patients with eccentric oesophagus under general anaesthesia. We use ultrasound to determined the position of the oesophagus after patient under general anaethesia ( to group them under central oesophagus and eccentric oesophagus) and also to determine the success of oesophagus occlusion.

SECONDARY OUTCOMES:
The number of patients with central oesophagus under general anesthesia, successfully occluded by using cricoid pressure. | ultrasound assessment of oesophagus done after general anaesthesia and during application of cricoid pressure
  The objective is to study the effectiveness of cricoid pressure in those patients with central oesophagus under general anaesthesia. We use ultrasound to determined the position of the oesophagus after patient under general anaethesia, and also to determine the success of oesophagus occlusion.

OTHER OUTCOMES:
incidence of variation of oesophagus position before and after general anaesthesia | ultrasound assessment of position of oesophagus before and after general anaesthesia
  We use ultrasound to determine the position of osephagus (central or eccentric) to determine the incidence of variation of oesophagus position before and after general anaesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Min Lim, M. Anaes, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee D, Czech AJ, Elriedy M, Nair A, El-Boghdadly K, Ahmad I. A multicentre prospective cohort study of the accuracy of conventional landmark technique for cricoid localisation using ultrasound scanning. Anaesthesia. 2018 Oct;73(10):1229-1234. doi: 10.1111/anae.14399. Epub 2018 Jul 25. PMID 30044502
- [Background] Rice MJ, Mancuso AA, Gibbs C, Morey TE, Gravenstein N, Deitte LA. Cricoid pressure results in compression of the postcricoid hypopharynx: the esophageal position is irrelevant. Anesth Analg. 2009 Nov;109(5):1546-52. doi: 10.1213/ane.0b013e3181b05404. PMID 19843793
- [Background] Andruszkiewicz P, Wojtczak J, Wroblewski L, Kaczor M, Sobczyk D, Kowalik I. Ultrasound evaluation of the impact of cricoid pressure versus novel 'paralaryngeal pressure' on anteroposterior oesophageal diameter. Anaesthesia. 2016 Sep;71(9):1024-9. doi: 10.1111/anae.13518. PMID 27523050
- [Background] Byas-Smith M, Prinsell JR Jr. Ultrasound-guided esophageal occlusion during rapid sequence induction. Can J Anaesth. 2013 Mar;60(3):327-8. doi: 10.1007/s12630-012-9847-9. Epub 2012 Dec 20. No abstract available. PMID 23263978
- [Background] Votruba J, Zemanova P, Lambert L, Vesela MM. The Role of Airway and Endobronchial Ultrasound in Perioperative Medicine. Biomed Res Int. 2015;2015:754626. doi: 10.1155/2015/754626. Epub 2015 Dec 14. PMID 26788507
- [Background] Bhatia N, Bhagat H, Sen I. Cricoid pressure: Where do we stand? J Anaesthesiol Clin Pharmacol. 2014 Jan;30(1):3-6. doi: 10.4103/0970-9185.125683. PMID 24574584
- [Background] Kei J, Utschig EE, van Tonder RJ. Using Ultrasonography to Assess the Effectiveness of Cricoid Pressure on Esophageal Compression. J Emerg Med. 2017 Aug;53(2):236-240. doi: 10.1016/j.jemermed.2017.04.025. Epub 2017 Jun 8. PMID 28602458
- [Background] Smith KJ, Dobranowski J, Yip G, Dauphin A, Choi PT. Cricoid pressure displaces the esophagus: an observational study using magnetic resonance imaging. Anesthesiology. 2003 Jul;99(1):60-4. doi: 10.1097/00000542-200307000-00013. PMID 12826843
- [Background] Smith KJ, Ladak S, Choi PT, Dobranowski J. The cricoid cartilage and the esophagus are not aligned in close to half of adult patients. Can J Anaesth. 2002 May;49(5):503-7. doi: 10.1007/BF03017931. PMID 11983669
- [Background] SELLICK BA. Cricoid pressure to control regurgitation of stomach contents during induction of anaesthesia. Lancet. 1961 Aug 19;2(7199):404-6. doi: 10.1016/s0140-6736(61)92485-0. No abstract available. PMID 13749923